CLINICAL TRIAL: NCT05278078
Title: Investigation of the Slimming Myokines as Biomarkers Potential for Some Gastrointestinal (GIS) and Urinarysystem (US) Cancers and on the Effects of Nutritional and Psychology of Concerned Patients
Brief Title: Slimming Myokines, Cancers,Nutritional and Psychology Support
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, diler us altay, assoc.prof, Ordu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: ORDU551
Record Dates: First submitted 2022-02-11; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Cancer
Keywords: cachexia; irisin; adropine; nutrition; psychology
MeSH Terms: conditions — Neoplasms; Cachexia | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: 1. st group of cancer patients given psychological support
  2. nd group of cancer patients given nutrition education
  3. rd group of cancer patients who received psychological support and nutrition education
  4. th group of cancer patients who will not receive any support
Who Masked: Participant
Masking Description: Participants in the study will not know which group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- psychological support (Other): Psychological support will be given to the experimental group.
  Interventions: Other: psychological support
- nutritional education (Other): Nutrition education will be given to the experimental group.
  Interventions: Other: nutritional education
- psychological support and nutritional education (Other): psychological support and nutritional education will be given to the experimental group.
  Interventions: Other: psychological support and nutritional education
- no intervation (Other): No intervention will be applied to the control group
  Interventions: Other: no intervation

INTERVENTIONS:
Other: psychological support — psychological support will be given to the patients in the experimental group.
  Other Names: experimental group.
  Arms: psychological support
Other: nutritional education — nutritional education will be given to the patients in the experimental group.
  Other Names: experimental group.
  Arms: nutritional education
Other: psychological support and nutritional education — psychological support and nutritional education will be given to the patients in the experimental group.
  Other Names: experimental group.
  Arms: psychological support and nutritional education
Other: no intervation — No intervention will be applied to the control group
  Other Names: control group
  Arms: no intervation

SUMMARY:
With the project investigators propose, investigators aim to find answers to the following questions: The fact that irisin and atropine are slimming the proteins that cause an increase in weight loss, and the excessive wasting (cachexia) in some types of cancer makes us wondering whether these factors may be cachectic factors for some GIS and US cancers? It is aimed to determine the relationship between irisin, atropine, some cachectic factors (PIF, ZAG), and cytokines (TNF-α, IL-1, IL-6) at tissue and plasma levels in these types of cancer. In addition, will psycho and nutrition education be applied to patients have an effect on cachexia? Experimental approaches to be used to find answers to such questions make this project unique.

DETAILED DESCRIPTION:
Cancer is the excessive and uncontrolled proliferation of a group of cells in the body. Problems experienced in cancers (cachectic cancers) which are known to be more underweight than other types of cancer; nutritional deficiencies, increasing muscle and adipose tissue atrophy, and psychological problems accompanying cachexia. Weight loss is approximately 60-80% in some GIS and US cancers. Although the mechanism of weight loss in cancer has not been fully elucidated, the importance of proinflammatory cytokines (Tumor necrosis faktör-α (TNF-α), Interleukin-1 (IL-1), Interleukin-6 (IL-6) factors over-synthesized by the body and factors causing muscle and fat atrophy (Proteolysis inducing factors (PIF)and Zinc- α-2 glycoprotein (ZAG) released from tumor cells, is known, but new and more precise agents for the treatment of cachexia are under investigation.

With the project investigators propose, investigators aim to find answers to the following questions: The fact that irisin and adropin are slimming the proteins that cause an increase in weight loss, and the excessive wasting (cachexia) in some types of cancer makes us wonder whether these factors may be cachectic factors for some GIS and US cancers? It is aimed to determine the relationship between irisin, atropine, some cachectic factors (PIF, ZAG), and cytokines (TNF-α, IL-1, IL-6) at tissue and plasma levels in these types of cancer. In addition, will psychoeducation and nutrition education be applied to patients have an effect on cachexia? Experimental approaches to be used to find answers to such questions make this project unique.

In this project, first of all, irisin and atropine will be compared to a combination of cachectic factors and cytokines due to, whether the effect of irisin and atropine on the formation of cancer cachexia at the level of gene and protein in tissue and plasma samples taken from 240 patients diagnosed with GIS (gastric, colon) and UC (bladder, renal) cancer. Nutritional and psychological education will be provided at regular intervals and the patient parameters will be remeasured at the plasma levels. In addition, body mass index monitoring and routine biochemical tests of all patients will be performed during this period. Statistically, Student-t will be used in binary comparisons and ANOVA tests will be used in triple comparisons.

If our hypothesis is realized, new cachectic factors have been identified, specific markers have been identified for GIS and UC cancers, the effect of psychological and nutritional education on cachexia will be answered within the scope of this project.

In line with the data to be obtained from this project in terms of career planning, atrophy and cachexia can be slowed down by injection of irisin and atropine to animals with cachectic cancer models in future projects and it can be planned to treat cancer types with high attenuation. In cancer patients, whose name creates fear in the society, affects people both physiologically and psychologically, and leads people to the bottom in the weakening coexistence, investigators aim to prevent psychological improvement as well as to prevent nutritional deficiencies and to increase the life expectancy in a lifetime. This multicenter and interdisciplinary project that investigators envisaged will enable us to show that investigators are ready for international projects.

ELIGIBILITY:
Inclusion Criteria:

Must be older than 18 years of age, Clinical diagnosis of pancreatic, colon, renal, bladder cancer, and not having any other chronic disease.

Exclusion Criteria:

* major gastrointestinal disease, chronic renal failure, uncontrolled diabetes, and HIV
* body mass index>30kg/m2,
* patients receiving drug therapy that modulates metabolism or weight deeply,

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Hospital-Anxiety Scale | 12 weeks
  The scale is applied to patients with physical illness and those applying to primary health care services. The scale consists of 14 questions in total. Seven of them (odd numbers) measure anxiety and the other seven (even numbers) measure depression. Scoring; Each item is scored differently. Items 1, 3, 5, 6, 8, 10, 11, and 13 show decreasing severity and the scoring is 3,2,1, 0. On the other hand, the 2nd, 4th, 7th, 9th, 12th, and 14th items are scored as 0,1,2,3. The total scores of the subscales are obtained by summing these item scores. While collecting the 1st, 3rd, 5th, 7th, 9th, 11th, and 13th items for the anxiety subscale; for depression subscale; The scores of the 2nd, 4th, 6th, 8th, 10th, 12th, and 14th items are added up. Interpretation; As a result of the study conducted in Turkey, the cut-off score for the anxiety subscale was found to be 10/11 and 7/8 for the depression subscale. Accordingly, those above these scores are considered at risk.
Holistic Well-being Scale | 12 Weeks
  Turkish validity and reliability were performed in 2019 in cancer patients. The scale is a 10-point Likert-type scale that measures holistic well-being with 30 items and 7 dimensions and is graded from completely disagree (1) to completely agree (10). Sub-dimensions of the scale: Non-attachment (18, 12, 24, 5, 25), distressing emotion (6, 21, 1, 28, 3), distressing perception (17, 8, 7, 29, 30), spiritual deterioration (20, 26, 2, 4), cognitive awareness (22, 13, 19, 11), general mood (15, 10, 14, 23), spiritual self-care (9, 16, 27). The 4th item in the scale is reverse coded. There is no cut-off point in the scale. The highest score that can be obtained from the scale is 300, and the lowest score is 30. Cronbach's alpha value ranged from 0.670 to 0.892.
Determination of slimming myokines, cachectic factors, cytokines protein levels by ELISA method | 12 weeks
  After reaching a sufficient number of patients, slimming myokines, cachectic factors, cytokines protein levels will be measured by the commercial kits ELISA (Enzyme-Linked Immunosorbent Assay) method.ELISA technique is the gold standard for quantitation of soluble proteins and provides rapid and consistent results that are easy to analyze.
Hemoglobin measurument in plasma samples | 12 weeks
  Hemoglobin (Hgb( g/dL); grams of hemoglobin per deciliter.
Body Mass Index Measurument | 12 weeks
  Especially body mass indexes of all patients weight and height will be combined to report BMI in kg/m^2 will be measured again at the beginning of the study and after the nutrition and psychological training.
C-reactive protein measurument in plasma samples | 12 weeks
  C-reactive protein (CRP(mg/L) milligrams of CRP per liter. It is possible to say that high CRP levels indicate an acute inflammatory reaction or an infection in the body, and a decrease in CRP levels indicates that the inflammatory reaction or infection has started to decrease
Aspartate transaminase measurument in plasma samples | 12 weeks
  Aspartate transaminase (AST(U/L) units of AST per liter.Plasma AST (aspartate transaminase) level is commonly measured clinically as a biomarker for liver health. The test is part of blood panels.
Alanine transaminase measurument in plasma samples | 12 weeks
  Alanine transaminase (ALT (U/L) units of ALT per liter. Plasma ALT level is commonly measured clinically as a biomarker for liver health. The test is part of blood panels.
Urea measurument in plasma samples | 12 weeks
  Urea (mg/dL)milligrams of urea per deciliter. Blood urea nitrogen (BUN) is a medical test that measures the amount of urea nitrogen found in the blood. The liver produces urea in the urea cycle as a waste product of the digestion of protein. Normal human adult blood should contain 6 to 20 mg/dL (2.1 to 7.1 mmol/L) of urea nitrogen.
total protein measurument in plasma samples | 12 weeks
  Total protein (g/dL) grams of total protein per deciliter. A total protein test is requested if you have a complaint about your nutritional status, such as weight loss. In the presence of symptoms suggestive of liver or kidney diseases or in the presence of symptoms such as fluid pooling (edema) in the tissues, it may be requested together with other tests.
Creatinine measurument in plasma samples | 12 weeks
  Creatinine(mg/dL) milligrams of creatinine per deciliter. Normal creatinine values average 0.6-1.3 mg/dL. If this value is above 2.0, renal failure is considered. However, in some cases, it has been observed that the creatinine value increases due to the rapid muscle metabolism in athletes who do heavy sports.
Cancer antigen 15-3 measurement in plasma samples | 12 weeks
  Cancer antigen 15-3 (CA15-3) (U/mL) units of CA 15-3 per milliliter. Cancer antigen 15-3 is a protein made by a variety of cells, particularly breast cancer cells. The protein moves into the blood, where it can be measured.CA15-3 levels are higher than normal in most women with breast cancer that has spread to other parts of the body (called metastatic breast cancer). Not all types of breast cancer will cause CA 15-3 levels to rise, as some types of cancer cells don't over-produce the antigen.
Cancer antigen 19-9 measurement in plasma samples | 12 weeks
  Cancer antigen 19-9 (U/mL) units of CA 19-9 per milliliter. This test measures the amount of a protein called CA 19-9 (cancer antigen 19-9) in the blood. CA 19-9 is a type of tumor marker. Tumor markers are substances made by cancer cells or by normal cells in response to cancer in the body.
Carcinoembryonic antigen (CEA) measurement in plasma samples | 12 weeks
  carcinoembryonic antigen (CEA)(ng/mL) nanograms of carcinoembryonic antigen per milliliter. Carcinoembryonic antigen (CEA) is a protein normally found in very low levels in the blood of adults. The CEA blood level may be increased in certain types of cancer and non-cancerous (benign) conditions. A CEA test is most commonly used for colorectal cancer.
RNA isolation from Tissue Samples | 12 weeks
  All tissue samples will be studied simultaneously by taking sections from the FFPE block.
  In our study, Invitrogen brand Pure Link to FFPE Total RNA isolation kit will be used. The operating procedure in the kit protocol will be followed. The spectrophotometric method will be used to determine the amount and quality of RNAs obtained before cDNA extraction.
  1 μl of the obtained RNAs will be loaded into the BioSpec-Nano (Shimadzu, Kyoto, Japan) device for contamination and concentration determination. The 260/280 absorbance ratio should ideally be around 2 for RNA samples. Samples that are too far from this value mean that there is contamination and RNA isolation will be repeated. RNA concentrations will be diluted to 100 μg/ml so that the initial RNA amounts of all samples are equal before cDNA translation.
cDNA extraction | 12 weeks
  ipsogen RT Kit (cDNA synthesis kit) will be used to convert the obtained Total RNA to cDNA. The operating procedure in the kit's protocol will be followed. The mixtures created will be exposed to 25°C for 10 minutes, 50°C for 60 minutes, 85°C for 5 minutes, and 4°C for 5 minutes within the reverse transcription (RT) program. cDNAs will be stored at -20°C until Real-Time PCR is performed. If necessary, it will be stored at -80oC to prolong the lifetime of cDNAs.
Expression analysis of slimming myokines, cachectic factors, cytokines genes by Real-Time PCR | 12 weeks
  The measurement of the slimming myokines, cachectic factors, cytokine parameters at the gene levels in the tissues is planned to be measured by the GeneaQ device will be used. The operating procedure in the kit's protocol will be followed.